CLINICAL TRIAL: NCT04244656
Title: A Phase 1 Dose Escalation and Cohort Expansion Study of the Safety and Efficacy of Anti-BCMA Allogeneic CRISPR-Cas9-Engineered T Cells (CTX120) in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: A Safety and Efficacy Study Evaluating CTX120 in Subjects With Relapsed or Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Patients to be followed up in the CRSP-ONC-LTF study
Sponsor: CRISPR Therapeutics AG (Industry)
Responsible Party: Sponsor
Organization: CRISPR Therapeutics (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CRSP-ONC-002
Record Dates: First submitted 2020-01-24; First posted 2020-01-28 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma
Keywords: CAR T; Allogeneic; Multiple myeloma; CRISPR-Cas9
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CTX120 (Experimental): Administered by IV infusion following lymphodepleting chemotherapy.
  Interventions: Biological: CTX120

INTERVENTIONS:
Biological: CTX120 — CTX120 B-cell maturation antigen (BCMA)-directed T-cell immunotherapy comprised of allogeneic T cells genetically modified ex vivo using CRISPR-Cas9 gene editing components.

SUMMARY:
This is a single-arm, open-label, multicenter, Phase 1 study evaluating the safety and efficacy of CTX120 in subjects with relapsed or refractory multiple myeloma.

ELIGIBILITY:
Key Inclusion Criteria:

1. Age ≥18 years.
2. Relapsed or refractory multiple myeloma, as defined by IMWG response criteria and treatment with at least 2 prior lines of therapy.
3. Eastern Cooperative Oncology Group performance status 0 or 1.
4. Adequate renal, liver, cardiac and pulmonary organ function
5. Female subjects of childbearing potential and male subjects must agree to use acceptable method(s) of contraception from enrollment through at least 12 months after CTX120 infusion.

Key Exclusion Criteria:

1. Prior allogeneic stem cell transplant (SCT).
2. Less than 60 days from autologous SCT at time of screening and with unresolved serious complications.
3. Prior treatment with any gene therapy or genetically modified cell therapy, including CAR T cells or natural killer cells, or BCMA-directed therapy.
4. Evidence of direct central nervous system (CNS) involvement by multiple myeloma.
5. History or presence of clinically relevant CNS pathology such as a seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, any autoimmune disease with CNS involvement.
6. Unstable angina, clinically significant arrhythmia, or myocardial infarction within 6 months of enrollment.
7. Active HIV, hepatitis B virus or hepatitis C virus infection.
8. Previous or concurrent malignancy, except basal cell or squamous cell skin carcinoma, adequately resected and in situ carcinoma of cervix, or a previous malignancy that was completely resected and has been in remission for ≥5 years.
9. Use of systemic anti-tumor therapy or investigational agent within 14 days prior to enrollment.
10. Primary immunodeficiency disorder or active autoimmune disease requiring steroids and/or other immunosuppressive therapy.
11. Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
Part A (dose escalation): Incidence of adverse events | From CTX120 infusion up to 28 days post-infusion
  Adverse events defined as dose-limiting toxicities
Part B (cohort expansion): Objective response rate | From CTX120 infusion up to 60 months post-infusion
  Objective response rate per International Myeloma Working Group (IMWG) response criteria.

SECONDARY OUTCOMES:
Progression Free Survival | From date of CTX120 infusion and date of disease progression or death due to any cause, assessed up to 60 months
Overall Survival | From date of CTX120 infusion until date of death due to any cause, assessed up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Annie Weaver, PhD, Study Director — CRISPR Therapeutics
Locations (10):
- United States (4):
  - University of Chicago, Chicago, Illinois
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
- Australia (2):
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- University Health Network, Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- Spain (3):
  - Institut Catala d'Oncologia Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario de Salamanca, Salamanca

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bruno B, Wasch R, Engelhardt M, Gay F, Giaccone L, D'Agostino M, Rodriguez-Lobato LG, Danhof S, Gagelmann N, Kroger N, Popat R, Van de Donk NWCJ, Terpos E, Dimopoulos MA, Sonneveld P, Einsele H, Boccadoro M. European Myeloma Network perspective on CAR T-Cell therapies for multiple myeloma. Haematologica. 2021 Aug 1;106(8):2054-2065. doi: 10.3324/haematol.2020.276402. PMID 33792221